CLINICAL TRIAL: NCT04595123
Title: Impact of COVID-19 Pandemic in Perinatal Mental Health
Brief Title: Impact of COVID-19 Pandemic in Perinatal Mental Health (RISEUP-PPD-COVID-19)
Status: Completed | Type: Observational
Sponsor: University of Minho (Other)
Collaborators: Universidad Loyola Andalucia (Other); Beder College University. Albania (Unknown); Mackenzie Presbiterian University, São Paulo, Brazil (Other); Medical University of Sofia (Other); European University Cyprus (Other); Groupe Hospitalier du Havre (Other); University of Athens (Other); Bar-Ilan University, Israel (Other); University of Malta (Other); Mount Carmel Health System (Other); University of Coimbra (Other); Universidade Católica Portuguesa (Other); Instituto de Saude Publica da Universidade do Porto (Other); University of Huelva (Other); Instituto de Investigação Biomédica de Malaga. Spain (Unknown); Universidad Nacional de Educación a Distancia (Other); Kırklareli University (Other); King's College London (Other); Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, Ana Mesquita, PhD, University of Minho
Other Study IDs: RISEUP-PPD-COVID-19
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Post Traumatic Stress Disorder; Depression; Anxiety; Psychological Distress
Keywords: Perinatal mental health; Women; Anxiety; Depression; COVID-19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Coronavirus disease 2019 (COVID-19) is a new pathology, declared a public health emergency by the World Health Organization, which can have negative consequences for pregnant women and their newborns. It is estimated that 1 in 5 women will develop a mental illness in the perinatal period. COVID-19 pandemic has been associated with anxiety and depression in the population. The current pandemic is a unique stressor with potentially wide-ranging consequences in the perinatal period, but little is known about the impact of COVID-19 on perinatal mental health. Thus, the objective of this study is to explore the experiences of pregnant and new mothers during the current pandemic, particularly its impact on perinatal mental health (including depression, anxiety, PTSD and psychological distress). Methods: The study design is a prospective observational study, with a baseline assessment and three follow-ups: one month; three months; and six months post baseline. This international study will be carried out in 11 European countries (Albania, Bulgaria, Cyprus, France, Greece, Israel, Malta, Portugal, Spain, Turkey, United Kingdom) Chile and Brazil. The study population will comprise pregnant women and new mothers with an infant under six months of age, covering a broad range of women across the perinatal period. Ethics and dissemination: The study and handling of the data will follow all national required data protection standards. Each researcher (or team of researchers) involved will submit the project to their local ethical committee before starting the project. Results from the project will be disseminated in peer reviewed journals and international conferences.

DETAILED DESCRIPTION:
This study is co-sponsored by University of Loyola, Seville, Spain and from University of Minho, Braga Portugal. Emma Motrico and Ana Mesquita as Principal Investigators of the study are the Responsible Parties.

Coronavirus disease 2019 (COVID-19) is a new pathology, declared a public health emergency by the World Health Organization that appeared more benign for pregnant women than for their newborns. COVID-19 pandemic is causing fear, anxiety and depression in the population. At the same time, pregnancy and postpartum is a period of increased risk for mental illness. It is estimated that 1 in 5 women will develop a mental illness in the perinatal period. Perinatal depression is the most common mental illness experienced during pregnancy and postpartum and has long-lasting adverse effects on women and their babies, bringing a strong burden to their families and society as a whole. The current COVID-19 pandemic is a unique stressor with potentially wide-ranging consequences in the perinatal period. Evidence coming from past epidemics, namely ZIKV infection (Zika virus) highlight the importance of examining mental health in light of stressful events experienced during pregnancy and the postpartum period and of long-term support for these mothers. There has been an increase in the prevalence of perinatal depression, anxiety and psychological distress after the announcement of the SARS-CoV-2 outbreak.

The project Research Innovation and Sustainable Pan-European Network in Peripartum Depression Disorder - Riseup-PPD" (CA18138) is a Cost Action (European Cooperation in Science and Technology) funded by the Horizon 2020 Framework Programme of the European Union. The project aims to establish a European multidisciplinary network of experts dedicated to the understanding of Peripartum Depression (PPD), from its prevention and assessment to its treatment and evaluation of impact, considering the women, the newborns and the wider family and social systems. Researchers from different core expertise (clinical medicine, psychology, health sciences, mathematic, media and communications) from 23 European countries and six international countries participate in the COST Action Riseup-PPD. In order to promote best practices in perinatal mental health that may mitigate the impact of COVID-19 management in women's mental health, the COST Action Riseup- PPD has decided to create a new Task Force "Perinatal Mental Health and COVID-19 pandemic". One of the main objectives of this crosscutting Task Force is to evaluate the impact of COVID-19 on perinatal mental health. Aims: Test the hypothesis that COVID-19 pandemic is associated with increased perinatal mental illness.

Methods Study design: Prospective observational study, with a baseline assessment and three follow-ups: one-month; three months; and six-months.

Setting: 11 European countries - Albania, Bulgaria, Cyprus, France, Greece, Israel, Malta, Portugal, Spain, Turkey, United Kingdom - Chile and Brazil. Participants: Pregnant women and new mothers with an infant under six months of age. Data from additional countries could also be include in the future to this study, if using the same instruments.

Study size: A representative sample was calculated according to number of newborns in the previous year in each country. The investigators estimate a minimum group size of 300 women per country. The estimation is based on an α-level of 0.05 and heterogeneity equal to 50%.

Variables and questionnaires Predictor variables/independent variables:

COVID-19 and Public health measures. Data on COVID-19 includes for each country (1) date of first confirmed case, (2) date of first death, and (3) at the date of questionnaire release: (3.1) number of confirmed cases, (3.2) number of recoveries (3.3) number of deaths. Data on public health measures adopted to contain the COVID-19 pandemic will include date and guidelines for (1) general restrictions (events, sports, religious ceremonies); (2) home confinement; (3) social distancing; (4) schools and services closing; and (5) restrictions to circulation within the country and between countries (including external border closure). Data on the deconfinement plan, including (1) general deconfinement (events, sports, religious ceremonies); (2) rules for circulating in public transport and services (including mandatory use of face masks); (3) schools reopening; and (4) services reopening.

Sociodemographic variables: date of birth, ethnicity, education, marital status, residence and questions about number of people living at home and numbers of weeks in confinement.

Coronavirus Perinatal Experiences Impact Survey (COPE-IS) - perinatal experiences; exposure and symptoms; financial impact; social support impact; social distancing and activity restriction; coping and adjustment; emotional impact; health background, mental health, and substance use.

In the follow-up assessments, experiences of new and expectant mothers will be measured with the Coronavirus Perinatal Experiences Scale-Impact Update (COPE-IU) and the Coronavirus Perinatal Experiences Scale - Care Follow Up (COPE-CF). The COPEIU evaluates exposure to COVID-19 and symptoms; impact on daily life, experiences, and feelings; the COPE-CF evaluates perceived support and care and the social and financial impact of the pandemic.

Perinatal experiences: Includes questions about if it is/was her first pregnancy, health problems during pregnancy, type of pregnancy, pre and postnatal care support, resources available from pre and postnatal care, changes experienced as a result of COVID-19 and question related to concerns about changes in family/friends support, medical care during the baby´s birth and child´s health as a result of the COVID-19 outbreak. Specifically, for women of a child younger than six months, this also includes other questions about city and place of birth, breastfeeding, changes experienced in birth plans and level of distress experienced related to changes in baby´s birth and postnatal experiences. Exposures and symptoms: Pregnant women/ new mothers and their family have been exposed to or are experiencing any symptoms like those seen in COVID-19. This includes questions about the diagnosis of COVID-19, symptoms compatible with coronavirus, contact with someone who has been diagnosed withCOVID-19, anyone close died due to COVID-19, and the degree of distress about COVID-19 related symptoms or potential illness. Financial impact: type of employment, impact of the pandemic on future employment and financial impact of the COVID-19 outbreak.

Social support impact: Support seeking, support provided, need for support, perceived support, and level of distress experienced with disruptions to social support due to the COVID-19 outbreak.

Coping and adjustment: Includes 23 coping strategies (problem-focused or emotion-focused) in response the stress related to the COVID-19 outbreak.

Emotional impact: Impact of COVID-19 on mental health - subjective impact of the COVID-19 outbreak on stress levels and mental health, sleep, and daily energy levels and the positive and negative impacts of the COVID-19 outbreak on daily life.

Health background, mental health, and substance use: Five mental health and substance use questions from the John's Hopkins COVID-19 Mental Health Measurement Working Group: 1) the woman's history of medical conditions; 2) household history of medical conditions; 3) current mental illness; 4) current substance use; and 5) treatment of medical conditions.

Psychological distress using the Brief Symptom Inventory-18 (BSI-18), omitting suicidality.

Dependent/outcome variables: Maternal and perinatal mental health outcomes will be evaluated - depression, anxiety and Posttraumatic Stress Disorder (PTSD), Measurements include the Edinburgh Postnatal Depression Scale (EPDS), the Generalized Anxiety Disorder Screener (GAD-7), a subset of 10 questions from the Posttraumatic Stress Disorder (PTSD) Checklist for DSM-5 related with COVID-19 included in COPE-IS and COPE-IU questionnaire [

(1) Feeling super alert or watchful or on guard; 2) Feeling jumpy or easily startled; 3) Having difficulty concentrating; 4) Trouble experiencing positive feelings; 5) Feeling guilty or blaming yourself; 6) Feeling irritable, angry or aggressive; 7) Repeated disturbing and unwanted thoughts about the COVID-19 outbreak; 8) Repeated disturbing dreams about the COVID-19 outbreak; 9) Trying to avoid information or reminders about the COVID-19 outbreak; and 10) Taking too many risks or doing things that could cause the participants harm]

Data collection: Participants will be recruited through social media (Twitter, WhatsApp, Facebook and Instagram, Reddit, Researchgate, Linkedin, Ya, etc.), networks of organizations (including universities, health centers, NGOs working on the field of perinatal mental health), policymakers, local organizations, and other stakeholders. Participants will also be recruited directly by message or email.

Participants are provided with a link to a digital survey that will direct them to an electronic consent form that provides an overview of what to expect and states that participation is voluntary, the purpose of research, possible risks, possible benefits, confidentiality protection, and appropriate alternatives. The baseline assessment is anticipated to be 20 minutes long. Eligible participants who complete the initial survey will be asked to participate in follow-up assessments.

Participation in the follow-ups will be optional and participants will have to provide their consent to be contacted by email or phone; attached to this request the investigators will provide a clear plan to protect confidentiality of information and contact information data protection plan (this will also be provided in the Informed Consent).

Ethical standards and safety monitoring: The study and handling of the data will follow all national required data protection standards. Each researcher (or team of researchers) involved will submit the project to local ethical committee before starting the project. Participants are provided with a link to an informed consent form before starting the study. If they agree to participate, only then will they proceed to the online survey. The consent form provides an overview of the aims of the study, what to expect and explains how confidentiality will be protected. Clarification of the voluntary nature of participation in the survey and of absence of compensation will be provided. Data should be collected anonymously, although email or/and phone number will be necessary for the follow-up assessments. Inclusion of vulnerable subjects is justified for this study because the purpose of the study is to examine pregnant or breastfeeding women. The research contains negligible risks as there is no more foreseeable risk of harm or discomfort other than potential inconvenience during participation. The study does not include deception, but some questions of the survey can elicit changes in the emotional state of participants. In order to address this issue, a debriefing procedure will be made available; at the end of the survey, information about resources in each country on mental health, perinatal care and COVID-19 as well as contacts of the research team will be given in case participants would like to have additional information. Information about the global results of the study will be provided upon request.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or biological mother of a child six months old or younger
* 18 years of age or older
* Live in one of the countries of the study
* Accept to participate in the study

Exclusion Criteria:

* Not pregnant and not biological mother of a child 6 months old or younger
* Younger than 18 years old
* Not live in one of the countries of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is pregnant women and new mothers with an infant under six months of age. The rationale is to evaluate during the six-month follow-up the "peripartum period", from pregnancy to one year following childbirth
Sampling Method: Non-Probability Sample
Enrollment: 7642 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | June 2020- June 2021
  Number of depressive symptoms evaluated by Edinburgh Postnatal Depression Scale (EPDS).
  Scores range from 0 to 30. Higher scores mean worse outcome
Posttraumatic Stress Disorder | June 2020- June 2021
  Number of Post-Traumatic Stress Disorders (PTSD) symptoms evaluated by check list of DSM-5. HIgher number of symptoms mean worse outcomes
Anxiety symptoms | June 2020- June 2021
  Number of anxiety symptoms evaluated by General Anxiety Disorder questionnaire (GAD 7). Scores range from 0 to 21. Higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Mesquita, PhD, Principal Investigator — University of Minho; Emma Motrico, PhD, Principal Investigator — Universidad Loyola Andalucia
Locations (13):
- Beder College University, Tirana, Albania
- Universidade Presbiteriana Mackenzie, São Paulo, Brazil
- Sofia University, Sofia, Bulgaria
- Universidad de Concepción, Concepción, Chile
- European University Cyprus, Nicosia, Cyprus
- Groupe Hospitalier du Havre, Le Havre, France
- University of Athens, Athens, Greece
- Bar-Ilan University, Ramat Gan, Israel
- University of Malta, Msida, Malta
- Universidade do Minho, Braga, Portugal
- Universidad Loyola Andalucia, Seville, Spain
- Kırklareli Üniversitesi, Kırklareli, Turkey (Türkiye)
- King'S College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu N, Li W, Kang Q, Xiong Z, Wang S, Lin X, Liu Y, Xiao J, Liu H, Deng D, Chen S, Zeng W, Feng L, Wu J. Clinical features and obstetric and neonatal outcomes of pregnant patients with COVID-19 in Wuhan, China: a retrospective, single-centre, descriptive study. Lancet Infect Dis. 2020 May;20(5):559-564. doi: 10.1016/S1473-3099(20)30176-6. Epub 2020 Mar 24. PMID 32220284
- [Background] World Health Organization (2020). WHO guidelines on Intrapartum care for a positive childbirth experience and Interim guidance on Clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected. https://www.who.int/docs/default-source/coronaviruse/clinical-management-of-novel-cov.pdf
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Fertility: Assessment and Treatment for People with Fertility Problems. London: Royal College of Obstetricians & Gynaecologists; 2013 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK247932/ PMID 25340218
- [Background] Hahn-Holbrook J, Cornwell-Hinrichs T, Anaya I. Economic and Health Predictors of National Postpartum Depression Prevalence: A Systematic Review, Meta-analysis, and Meta-Regression of 291 Studies from 56 Countries. Front Psychiatry. 2018 Feb 1;8:248. doi: 10.3389/fpsyt.2017.00248. eCollection 2017. PMID 29449816
- [Background] Shorey S, Chee CYI, Ng ED, Chan YH, Tam WWS, Chong YS. Prevalence and incidence of postpartum depression among healthy mothers: A systematic review and meta-analysis. J Psychiatr Res. 2018 Sep;104:235-248. doi: 10.1016/j.jpsychires.2018.08.001. Epub 2018 Aug 3. PMID 30114665
- [Background] Caparros-Gonzalez RA. [Maternal and neonatal consequences of coronavirus COVID-19 infection during pregnancy: a scoping review]. Rev Esp Salud Publica. 2020 Apr 17;94:e202004033. Spanish. PMID 32382001
- [Background] Moraes EV, Toledo OR, David FL, Godoi BN, Monteiro KA, Deluqui TC, Teixeira TW, Carvalho AL, Avelino MM. Implications of the clinical gestational diagnosis of ZIKV infection in the manifestation of symptoms of postpartum depression: a case-control study. BMC Psychiatry. 2019 Jun 26;19(1):199. doi: 10.1186/s12888-019-2157-9. PMID 31242891
- [Background] Dos Santos Oliveira SJG, Dos Reis CL, Cipolotti R, Gurgel RQ, Santos VS, Martins-Filho PRS. Anxiety, depression, and quality of life in mothers of newborns with microcephaly and presumed congenital Zika virus infection: a follow-up study during the first year after birth. Arch Womens Ment Health. 2017 Jun;20(3):473-475. doi: 10.1007/s00737-017-0724-y. Epub 2017 Apr 21. No abstract available. PMID 28429099
- [Background] Lebel C, MacKinnon A, Bagshawe M, Tomfohr-Madsen L, Giesbrecht G. Elevated depression and anxiety symptoms among pregnant individuals during the COVID-19 pandemic. J Affect Disord. 2020 Dec 1;277:5-13. doi: 10.1016/j.jad.2020.07.126. Epub 2020 Aug 1. PMID 32777604
- [Background] Wu, Y. T., Zhang, C., Liu, H., Duan, C. C., Li, C., Fan, J. X., ... & Guo, Y. (2020). Perinatal Depression of Women Along with 2019 Novel Coronavirus Breakout in China. Available at SSRN: https://ssrn.com/abstract=3539359 or http://dx.doi.org/10.2139/ssrn.3539359
- [Background] Thomason, M.E., Graham, A., VanTieghem, M.R. (2020). The COPE-IS: Coronavirus Perinatal Experiences - Impact Survey. Available on the Open Science Framework (OSF) at https://osf.io/uqhcv/.
- [Background] Thomason, M.E., Graham, A., Smyser, C.D., Rogers, C.E. (2020). The COPE-IU: Coronavirus Perinatal Experiences - Impact Update. Available on the Open Science Framework (OSF) at https://osf.io/uqhcv/
- [Background] Derogatis, L.R.(1993). BSI Brief Symptom Inventory: Administration, Scoring, and Procedure Manual (4th Ed.). Minneapolis, MN: National Computer Systems
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The PTSD Checklist for DSM-5 (PCL-5) - Extended Criterion A [Measurement instrument]. Available from https://www.ptsd.va.gov/
- [Background] Bracken-Roche D, Bell E, Macdonald ME, Racine E. The concept of 'vulnerability' in research ethics: an in-depth analysis of policies and guidelines. Health Res Policy Syst. 2017 Feb 7;15(1):8. doi: 10.1186/s12961-016-0164-6. PMID 28173859
- [Derived] Mesquita A, Costa R, Dikmen-Yildiz P, Faria S, Silvestrini G, Mateus V, Vousoura E, Wilson CA, Felice E, Ajaz E, Hadjigeorgiou E, Hancheva C, Contreras-Garcia Y, Dominguez-Salas S, Motrico E, Soares I, Ayers S. Changes to women's childbirth plans during the COVID-19 pandemic and posttraumatic stress symptoms: a cross-national study. Arch Womens Ment Health. 2024 Jun;27(3):393-403. doi: 10.1007/s00737-023-01403-3. Epub 2023 Dec 16. PMID 38102527
- [Derived] Mesquita A, Costa R, Bina R, Cadarso-Suarez C, Gude F, Diaz-Louzao C, Dikmen-Yildiz P, Osorio A, Mateus V, Dominguez-Salas S, Vousoura E, Levy D, Alfayumi-Zeadna S, Wilson CA, Contreras-Garcia Y, Carrasco-Portino M, Saldivia S, Christoforou A, Hadjigeorgiou E, Felice E, Buhagiar R, Hancheva C, Ajaz E, Uka A, Motrico E. A cross-country study on the impact of governmental responses to the COVID-19 pandemic on perinatal mental health. Sci Rep. 2023 Feb 16;13(1):2805. doi: 10.1038/s41598-023-29300-w. PMID 36797263
- [Derived] Motrico E, Galan-Luque T, Rodriguez-Dominguez C, Gomez-Gomez I, Dominguez-Salas S. Factors Associated with Post-Traumatic Stress Symptoms in Pregnant and Postpartum Women. J Womens Health (Larchmt). 2023 May;32(5):583-591. doi: 10.1089/jwh.2022.0400. Epub 2023 Feb 14. PMID 36787455
- [Derived] Wilson CA, Gomez-Gomez I, Parsons J, Costa R, Mesquita A, Vousoura E, Contreras-Garcia Y, Levy D, Mateus V, Christoforou A, Felice E, Dikmen-Yildiz P, Dominguez-Salas S, Motrico E. The Mental Health of Women with Gestational Diabetes During the COVID-19 Pandemic: An International Cross-Sectional Survey. J Womens Health (Larchmt). 2022 Sep;31(9):1232-1240. doi: 10.1089/jwh.2021.0584. Epub 2022 Jul 19. PMID 35856836
- [Derived] Gomez-Baya D, Gomez-Gomez I, Dominguez-Salas S, Rodriguez-Dominguez C, Motrico E. The influence of lifestyles to cope with stress over mental health in pregnant and postpartum women during the COVID-19 pandemic. Curr Psychol. 2022 Jun 15:1-20. doi: 10.1007/s12144-022-03287-5. Online ahead of print. PMID 35729900
- [Derived] Motrico E, Bina R, Dominguez-Salas S, Mateus V, Contreras-Garcia Y, Carrasco-Portino M, Ajaz E, Apter G, Christoforou A, Dikmen-Yildiz P, Felice E, Hancheva C, Vousoura E, Wilson CA, Buhagiar R, Cadarso-Suarez C, Costa R, Devouche E, Ganho-Avila A, Gomez-Baya D, Gude F, Hadjigeorgiou E, Levy D, Osorio A, Rodriguez MF, Saldivia S, Gonzalez MF, Mattioli M, Mesquita A; Riseup-PPD-COVID-19 Group. Impact of the Covid-19 pandemic on perinatal mental health (Riseup-PPD-COVID-19): protocol for an international prospective cohort study. BMC Public Health. 2021 Feb 17;21(1):368. doi: 10.1186/s12889-021-10330-w. PMID 33596889
- See also: Website of the project — https://momsduringcovid.org